CLINICAL TRIAL: NCT06278532
Title: Validation of the Lithuanian Version of the Brief Negative Symptoms Scale, Calgary Depression Scale for Schizophrenia, and the Schizophrenia Cognition Rating Scale
Brief Title: Validation of the Lithuanian Version of the BNSS, CDSS, and the SCoRS
Status: Recruiting | Type: Observational
Sponsor: Lithuanian University of Health Sciences (Other)
Responsible Party: Principal Investigator, Virginija Adomaitienė, Head of Psychiatry Department, Lithuanian University of Health Sciences
Other Study IDs: NEGKOG
Record Dates: First submitted 2024-01-16; First posted 2024-02-26 (Actual); Last update posted 2024-02-26 (Actual); Status verified 2024-02

CONDITIONS: Schizophrenia; Negative Symptoms in Schizophrenia; Depressive Symptoms Due to Primary Psychotic Disorder (Diagnosis); Cognitive Deficit
Keywords: Schizophrenia, Negative symptoms, Depressive symptoms of Schizophrenia, Cognitive deficits of Schizophrenia
MeSH Terms: conditions — Schizophrenia; Disease; Cognition Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Brief Negative Symptoms Scale — The Lithuanian Brief Negative Symptoms scale (BNSS) version will be used and validated. BNSS is used as a modern tool for the evaluation of negative symptoms of schizophrenia. Older tools used for negative symptoms evaluation often include symptoms from other dimensions of symptoms of schizophrenia, and BNSS evaluates negative symptoms specifically. BNSS is a semi-structured interview made of 13 items. There are six subscales: anhedonia (3 items), lack of normal distress (1 item), asociality (2 items), avolition (2 items), blunted affect (3 items) and alogia (2 items).
  Other Names: BNSS
Diagnostic Test: The Calgary Depression Scale for Schizophrenia — The Lithuanian version of the CDSS will be used and validated. CDSS is a tool used to evaluate depressive symptoms, specifically for patients with schizophrenia. Often, distinguishing between depressive and negative symptoms of schizophrenia is difficult. Therefore, it is recommended to use tools designed specifically for patients with schizophrenia. CDSS is the only depression scale designed to assess depression in people with a schizophrenia syndrome disorder. It is a semi-structured interview consisting of 9 items.
  Other Names: CDSS
Diagnostic Test: The Schizophrenia Cognition Rating Scale — The Lithuanian version of the SCoRS will be used and validated. SCoRS is a 20-item interview-based assessment tool that evaluates cognitive deficits and the degree to which these deficits impair specifically in patients with schizophrenia.
  Other Names: SCoRS

SUMMARY:
This study aims to validate the Lithuanian version of the Brief Negative Symptoms Scale, Calgary Depression Scale for Schizophrenia, and Schizophrenia Cognition Rating Scale in a Lithuanian sample. This will be done by comparing results obtained from the Brief Negative Symptoms Scale, Calgary Depression Scale for Schizophrenia, and Schizophrenia Cognition Rating Scale with results obtained from the Positive and Negative Symptoms Scale, the Montgomery Asberg Depression Rating Scale, and the Montreal Cognitive Assessment test.

DETAILED DESCRIPTION:
This scale validation study aims to validate the Lithuanian version of the Brief Negative Symptoms Scale, Calgary Depression Scale for Schizophrenia, and Schizophrenia Cognition Rating Scale Schizophrenia Cognition Rating Scale in the Lithuanian sample. The main aim of this study is:

• to evaluate the convergent and discriminant validity of Lithuanian versions of the Brief Negative Symptoms Scale, Calgary Depression Scale for Schizophrenia, and Schizophrenia Cognition Rating Scale.

Participants will be evaluated using the Positive and Negative Symptoms Scale (PANSS), Montgomery Asberg Depression Rating Scale (MADRS), Montreal Cognitive Assessment (MoCA) test, Brief Negative Symptoms Scale, Calgary Depression Scale for Schizophrenia, and Schizophrenia Cognition Rating Scale.

To discern the discriminant validity of the Brief Negative Symptoms Scale for negative symptoms, results from the Brief Negative Symptoms Scale will be compared to results from the positive and general subscale of the Positive and Negative Symptoms Scale and the Montgomery Asperger Depression Rating Scale. To discern the convergent validity of the Brief Negative Symptoms Scale for negative symptoms, results from the Brief Negative Symptoms Scale will be compared to the results from the negative subscale of the Positive and Negative Symptoms Scale and the Self-evaluation of Negative Symptoms scale.

To discern the discriminant validity of the Calgary Depression Scale for Schizophrenia for depressive symptoms of schizophrenia, results obtained from the Calgary Depression Scale for Schizophrenia will be compared to results obtained from the Positive and Negative Symptoms Scale and the Self-evaluation of Negative Symptoms scale. To check the convergent validity of the Calgary Depression Scale for Schizophrenia, results obtained from the Calgary Depression Scale for Schizophrenia will be compared to results obtained from the Montgomery Asperger Depression Rating Scale.

Finally, to check the discriminant validity of the Schizophrenia Cognition Rating Scale, results obtained from the Schizophrenia Cognition Rating Scale will be compared to results obtained from the Montgomery Asperger Depression Rating Scale and the Positive and Negative Symptoms Scale. In contrast, to prevent convergent validity, results obtained from the Schizophrenia Cognition Rating Scale will be compared to results obtained from the Montreal Cognitive Assessment test.

ELIGIBILITY:
Inclusion Criteria:

* age 18 - 65 years old;
* Diagnosis of F20, F25 or F21 according to ICD-10;
* Signed informed consent form.

Exclusion Criteria:

* Age younger than 18 or older than 65 years old;
* Did not sign the informed consent form;
* Legally inactive person
* Patients with a comorbid or primary diagnosis of mental retardation according to ICD-10 (F70 - F79);
* Patients with a comorbid or primary diagnosis of mental and behavioural disorders due to psychoactive substance use (F10 - F19)
* Patients with a comorbid of primary diagnosis of organic, including symptomatic, mental disorders (F00 - F09)

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Inpatients between 18 and 65 years old with a diagnosis of F20, F25, or F21, according to ICD-10, who sign the informed consent form and do not have any exclusion criteria, will be included in the study. We will not devide patients who have active psychotic symptoms and those who do not.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-12-11 (Actual); Primary Completion 2026-12-11 (Estimated); Study Completion 2026-12-11 (Estimated)

PRIMARY OUTCOMES:
Validated Lithuanian version of the Brief Negative Symptoms Scale. | Day 1
  Patients will be evaluated using the Lithuanian version of the Brief Negative Symptoms Scale (score 0 - 78; a greater score means more pronounced negative symptoms) once during the inpatient treatment. The results will be compared with the Positive and Negative Symptoms Scale score (0 - 210; a greater score means more pronounced symptoms of schizophrenia), Montgomery Asperger Depression Scale (Score 0 - 60; a greater score means greater symptoms of depression), Self-evaluation of Negative Symptoms Scale (score 0 - 40; greater score means more pronounced negative symptoms), and Montreal Cognitive Assessment Test (score 0 - 31; a greater score means better cognitive functions). Convergent and divergent validities will be calculated for each validated instrument by calculating correlations.
Validated Lithuanian version of the Calgary Depression Scale for Schizophrenia. | Day 1
  Patients will be evaluated using the Lithuanian version of the Calgary Depression Scale for Schizophrenia (score 0 - 27; a greater score means greater depression) once during the inpatient treatment, and the results will be compared with results from the Positive and Negative Symptoms Scale (score 0 - 210, greater score means more pronounced symptoms of schizophrenia), Montgomery Asperger Depression Scale (Score 0 - 60; greater score means greater symptoms of depression), and Self-evaluation of Negative Symptoms Scale (score 0 - 40; greater score means more pronounced negative symptoms). Convergent and divergent validities will be calculated for each validated instrument by calculating correlations.
Validated Lithuanian version of the Schizophrenia Cognition Rating Scale. | Day 1
  Patients will be evaluated using the Lithuanian version of the Schizophrenia Cognition Rating Scale (score 0 - 80; a greater score means worse cognitive functions; global functioning score 1 - 10 with a greater score meaning worse functioning) once during the inpatient treatment, and the results will be compared with results from the Montreal Cognitive Assessment Test (score 0 - 31; a greater score means better cognitive functions). Convergent and divergent validities will be calculated for each validated instrument by calculating correlations.

SECONDARY OUTCOMES:
Correlation between negative symptoms and cognitive deficits of schizophrenia | Day 1
  Correlation between negative symptoms evaluated with second-generation negative symptoms assessment tools (Brief Negative Symptoms Scale (score 0 - 78; a greater score means more pronounced negative symptoms) and Self-evaluation of Negative Symptoms scale (score 0 - 40; greater score means more pronounced negative symptoms) and Schizophrenia Cognition Rating Scale (score 0 - 80; a greater score means worse cognitive functions; global functioning score 1 - 10 with a greater score meaning worse functioning). Correlations between specific subscales of the Brief Negative Symptoms Scale, the Self-evaluation of Negative Symptoms Scale, and the Schizophrenia Cognition Rating Scale will be calculated. We will check for differences in correlation between different ages, education, duration of disease groups, and sexes.
Correlation between depressive symptoms and cognitive deficits of schizophrenia | Day 1
  Correlation between depressive symptoms evaluated with the Calgary Depression Scale for Schizophrenia (score 0 - 27; a greater score means greater depression) and Schizophrenia Cognition Rating Scale (score 0 - 80; a greater score means worse cognitive functions; global functioning score 1 - 10 with a greater score meaning worse functioning). Correlations between specific items of the Calgary Depression Scale for Schizophrenia and the Schizophrenia Cognition Rating Scale will be calculated. We will check for differences in correlation between different ages, education, duration of disease groups, and sexes.
Correlation between negative symptoms, cognitive deficits, depressive symptoms of schizophrenia and health-related quality of life | Day 1
  Correlation between results obtained from the Brief Negative Symptoms Scale score 0 - 78; a greater score means more pronounced negative symptoms), Self-evaluation of Negative Symptoms Scale (score 0 - 40; a greater score means more pronounced negative symptoms), Calgary Depression Scale for Schizophrenia (score 0 - 27; a greater score means greater depression), and the Schizophrenia Cognition Rating Scale (score 0 - 80; a greater score means worse cognitive functions; global functioning score 1 - 10 with a greater score meaning worse functioning) with results about the health-related quality of life of patients with schizophrenia evaluated with the 36-Item Short Form Survey (8 subscores scored from 0 percent to 100 percent, with more percents meaning better health-related quality of life) will be calculated. We will check for differences in correlation between different ages, education, duration of disease groups, and sexes.

CONTACTS AND LOCATIONS:
Overall Officials: Virginija Adomaitienė, Prof., Principal Investigator — Lithuanian University of Health Sciences
Locations (2):
- Lithuania (2):
  - Lithuanian University of Health Sciences Hospital Kaunas Clinics, Kaunas
  - Jonas Montvidas, Kaunas

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kirkpatrick B, Strauss GP, Nguyen L, Fischer BA, Daniel DG, Cienfuegos A, Marder SR. The brief negative symptom scale: psychometric properties. Schizophr Bull. 2011 Mar;37(2):300-5. doi: 10.1093/schbul/sbq059. Epub 2010 Jun 17. PMID 20558531
- [Background] Keefe RS, Davis VG, Spagnola NB, Hilt D, Dgetluck N, Ruse S, Patterson TD, Narasimhan M, Harvey PD. Reliability, validity and treatment sensitivity of the Schizophrenia Cognition Rating Scale. Eur Neuropsychopharmacol. 2015 Feb;25(2):176-84. doi: 10.1016/j.euroneuro.2014.06.009. Epub 2014 Jun 28. PMID 25028065
- [Background] Muller MJ, Brening H, Gensch C, Klinga J, Kienzle B, Muller KM. The Calgary Depression Rating Scale for schizophrenia in a healthy control group: psychometric properties and reference values. J Affect Disord. 2005 Sep;88(1):69-74. doi: 10.1016/j.jad.2005.04.005. PMID 16040126